CLINICAL TRIAL: NCT03198663
Title: POSSE Project: A Community-Level Intervention for Black YMSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Sybil Hosek, Clinical Psychologist, Cook County Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH104106 (NIH)
Record Dates: First submitted 2017-03-07; First posted 2017-06-26 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: HIV/AIDS and Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POSSE Intervention (Experimental)
  Interventions: Behavioral: POSSE
- Control (Other): Delayed intervention
  Interventions: Behavioral: POSSE

INTERVENTIONS:
Behavioral: POSSE — Popular-opinion leader

SUMMARY:
Black young men who have sex with men (BYMSM) are at high risk for contracting and transmitting HIV, and represent a priority population for developing effective interventions. Within the House Ball community (HBC), a clandestine subculture of the Black gay community, HIV is highly stigmatized. This stigma, coupled with high HIV prevalence rates and elevated levels of undiagnosed/untreated HIV infection, places BYMSM in HBCs at incredible risk for HIV infection. Community-level interventions that target social norms, behavior, and stigma in the HBC are sorely needed in order to make a broader impact among BYMSM. Building on prior work in the community, this study proposes to launch an innovative Effectiveness-Implementation Hybrid Type 2 trial to examine the effectiveness and implementation of a community-level HIV prevention intervention (called POSSE) based on popular opinion leader (POL) models across two cities with similar HBCs, Chicago and Philadelphia. The proposed study has two specific aims: 1) To determine the effectiveness of a POL intervention, POSSE, to decrease sexual risk behavior (UAI), STIs and HIV stigma among BYMSM in the HBC; and 2) To evaluate the processes, strategies, barriers and facilitators for the implementation of POSSE delivered across two distinct metropolitan areas with high HIV prevalence among BYMSM and similar House Ball Communities. To examine these aims, the investigators will first use social network strategies to identify, screen, and recruit POLs (n=75) from the Philadelphia HBC. The investigators will then gather baseline behavioral and biological (HIV/STI testing) data in both Chicago and Philadelphia (n=100 BYMSM per city) and train the Philadelphia POLs to implement the POSSE intervention. The investigators will conduct an implementation-focused process evaluation to assess fidelity to the POSSE intervention; number, content, spread, and acceptability of risk reduction messages; age appropriateness of the messages; acceptability of the overall intervention; and barriers/facilitators to implementation. Next, the investigators will complete follow-up assessments every 6 months post- intervention in both cities (n=100 BYMSM per city at each assessment point). The investigators will also assess behavior change in those delivering the intervention (POLs) at each assessment point. The investigators will conduct implementation-focused qualitative interviews with POLs (n=15) and community participants (n=30) from Philadelphia. Last, the investigators will implement POSSE in Chicago by repeating the steps outlined above, continuing assessments in both cities, and conducting qualitative interviews in Chicago.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Black,
* between the ages of 15 - 24 (inclusive), and
* in attendance at a HBC event at the time of the assessment.

Exclusion Criteria:

* intoxicated or otherwise unable to consent at time of enrollment

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1037 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
HIV incidence | 24 months

SECONDARY OUTCOMES:
STI incidence | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chicago, Illinois
  - Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No